CLINICAL TRIAL: NCT00354835
Title: Randomized Study of Vincristine, Dactinomycin and Cyclophosphamide (VAC) Versus VAC Alternating With Vincristine and Irinotecan (VI) for Patients With Intermediate-Risk Rhabdomyosarcoma (RMS)
Brief Title: Combination Chemotherapy and Radiation Therapy in Treating Patients With Newly Diagnosed Rhabdomyosarcoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARST0531; NCI-2009-00427 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 07-497; CDR0000487560; COG-ARST0531; ARST0531 (Other: Children's Oncology Group); ARST0531 (Other: CTEP); U10CA180886 (NIH); U10CA098543 (NIH)
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Results first posted 2017-07-25 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Adult Rhabdomyosarcoma; Childhood Alveolar Rhabdomyosarcoma; Childhood Botryoid-Type Embryonal Rhabdomyosarcoma; Childhood Embryonal Rhabdomyosarcoma; Localized Childhood Soft Tissue Sarcoma; Rhabdomyosarcoma; Sarcoma; Stage I Adult Soft Tissue Sarcoma AJCC v7; Stage II Adult Soft Tissue Sarcoma AJCC v7; Stage III Adult Soft Tissue Sarcoma AJCC v7
MeSH Terms: conditions — Rhabdomyosarcoma; Sarcoma | interventions — Cyclophosphamide; Dactinomycin; Irinotecan; Radiotherapy; Radiation; Vincristine

ARMS (2):
- Arm I (chemotherapy, radiotherapy) (Active Comparator): Patients receive VAC chemotherapy comprising vincristine IV over 1 minute on day 1 of weeks 1-13, 16, 19-25, 28, 31-37, and 40; dactinomycin IV over 1-5 minutes on day 1 of weeks 1, 4, 13, 16, 19, 22, 25, 28, 31, 34, 37,and 40; and cyclophosphamide IV over 1 hour on day 1 of weeks 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 31, 34, 37, and 40. Patients may also undergo radiotherapy 5 days a week for 4-6 weeks beginning in week 4.
  Interventions: Drug: Cyclophosphamide; Biological: Dactinomycin; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration; Radiation: Radiation Therapy; Drug: Vincristine Sulfate
- Arm II (chemotherapy, radiotherapy) (Experimental): Patients receive VAC chemotherapy alternating with VI chemotherapy comprising vincristine IV over 1 minute on day 1 of weeks 1-13, 16, 17, 19, 20, 22-26, 28, 31-34, 37, 38, and 40; dactinomycin IV over 1-5 minutes on day 1 of weeks 1, 13, 22, 28, 34, and 40; cyclophosphamide IV over 1 hour on day 1 of weeks 1,10, 13, 22, 28, 34, and 40; and irinotecan hydrochloride IV over 1 hour on days 1-5 of weeks 4, 7, 16, 19, 25, 31, and 37. Patients may also undergo radiotherapy 5 days a week for 4-6 weeks beginning in week 4.
  Interventions: Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Irinotecan Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration; Radiation: Radiation Therapy; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Biological: Dactinomycin — Given IV
  Other Names: Actinomycin A IV; Actinomycin C1; Actinomycin D; Actinomycin I1; Actinomycin IV; Actinomycin X 1; Actinomycin-[thr-val-pro-sar-meval]; Cosmegen; DACT; Dactinomycine; Lyovac Cosmegen; Meractinomycin
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; Irinomedac; Irinotecan Hydrochloride Trihydrate; Irinotecan Monohydrochloride Trihydrate; U-101440E
  Arms: Arm II (chemotherapy, radiotherapy)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Undergo radiotherapy
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This randomized phase III trial is studying two different combination chemotherapy regimens to compare how well they work when given together with radiation therapy in treating patients with newly diagnosed rhabdomyosarcoma. Drugs used in chemotherapy, such as vincristine sulfate, dactinomycin, cyclophosphamide, and irinotecan hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving combination chemotherapy together with radiation therapy may kill more tumor cells. It is not yet known which combination chemotherapy regimen is more effective when given together with radiation therapy in treating patients with rhabdomyosarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the early response rates, failure-free survival (FFS), and survival of patients with intermediate-risk rhabdomyosarcoma (RMS) treated with surgery, radiotherapy, and vincristine (vincristine sulfate), dactinomycin and cyclophosphamide (VAC) or VAC alternating with vincristine, irinotecan (irinotecan hydrochloride) (VI).

SECONDARY OBJECTIVES:

I. To compare FFS, local control, and survival of patients with intermediate-risk RMS treated with VAC and early (week 4) radiotherapy vs delayed (week 10) radiotherapy, using data from Intergroup Rhabdomyosarcoma Study (IRS)-IV for historic comparison.

II. To compare the acute and late effects of VAC to VAC alternating with VI, including the toxicity associated with concurrent VI and radiotherapy.

III. To compare the acute and late effects of VAC as delivered on this study to D9803 VAC.

IV. To correlate change in fludeoxyglucose F-18 positron emission tomography (FDG-PET) maximum standard uptake value (SUVmax) from week 1 to week 4 and 15 with FFS.

V. For VI treated patients, to correlate patient UDP glucuronosyltransferase 1 family, polypeptide A1 (UGT1A1) genotype with VI toxicity. VI. To correlate cytochrome P450, family 2, subfamily B, polypeptide 6 (CYP2B6), cytochrome P450, family 2, subfamily C, polypeptide 9 (CYP2C9), and glutathione S-transferase alpha 1 (GSTA1) genotypes with VAC toxicity.

VII. To prospectively evaluate and validate gene expression values with the intent to define the best diagnostic predictors and more powerful prognostic classifiers.

VIII. To assess the frequency of bladder dysfunction in patients with bladder, prostate, and pelvic sites of RMS 3-6 years after study enrollment.

OUTLINE: Patients are randomized to 1 of 2 treatment arms within 42 days of initial surgery or biopsy.

ARM I (VAC): Patients receive VAC chemotherapy comprising vincristine sulfate IV over 1 minute on day 1 of weeks 1-13, 16, 19-25, 28, 31-37, and 40; dactinomycin IV over 1-5 minutes on day 1 of weeks 1, 4, 13, 16, 19, 22, 25, 28, 31, 34, 37, and 40; and cyclophosphamide IV over 1 hour on day 1 of weeks 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 31, 34, 37, and 40.

ARM II (VAC/VI): Patients receive VAC chemotherapy alternating with VI chemotherapy comprising vincristine sulfate IV over 1 minute on day 1 of weeks 1-13,16, 17, 19, 20, 22-26, 28, 31-34, 37, 38, and 40; dactinomycin IV over 1-5 minutes on day 1 of weeks 1,13, 22, 28, 34, and 40; cyclophosphamide IV over 1 hour on day 1 of weeks 1,10, 13, 22, 28, 34, and 40; and irinotecan hydrochloride IV over 90 minutes on days 1-5 of weeks 4, 7, 16, 19, 25, 31, and 37.

In both arms, treatment continues in the absence of disease progression or unacceptable toxicity. Patients* in both arms also undergo radiotherapy 5 days a week for 4-6 weeks beginning in week 4 (except patients with alveolar RMS rendered group I by amputation OR patients needing week 1 emergency radiotherapy for symptomatic spinal cord compression).

NOTE: *Individualized local control plan that deviates from protocol-mandated radiotherapy allowed for patients =< 24 months of age.

After completion of study treatment, patients are followed up every 2-4 months for 4 years and then annually for 5-10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed embryonal RMS, botryoid or spindle cell variants of embryonal RMS, ectomesenchymoma, or alveolar RMS are eligible for this study
* Enrollment on COG-D9902 to confirm local histologic diagnosis with central pathology review is required for all patients
* Patients may be enrolled on ARST0531 and start protocol treatment prior to receipt of central pathology review results
* Patient must have Intermediate-risk RMS defined as:

  * Embryonal, botryoid, or spindle cell RMS, or ectomesenchymoma: stage 2 or 3 and group III OR
  * Alveolar RMS: stage 1-3 and group I-III
* Staging ipsilateral retroperitoneal lymph node dissection (SIRLND) is required for all patients >= 10 years of age with paratesticular tumors and for patients < 10 years with clinically or radiographically involved lymph nodes (except when extensive lymph node involvement, defined as two or more lymph nodes > 2 cm in dimension, is identified by imaging studies)
* Regional lymph node sampling or sentinel lymph node procedure is required for histologic evaluation in patients with extremity tumors
* Clinically or radiographically enlarged nodes should be sampled for histologic evaluation
* Detection of metastasis by optional FDG PET (not required for study enrollment); FDG PET may detect abnormalities suggestive of metastasis not identified by bone scan, computed tomography (CT), or bone marrow aspiration/biopsy; the prognostic significance of FDG PET-detected abnormalities is not clear; FDG PET-detected abnormalities MUST be confirmed to be metastases by an additional imaging modality (such as magnetic resonance imaging [MRI] or CT) OR pathologic confirmation; unless FDG PET abnormalities are confirmed by another imaging modality or biopsy, FDG PET abnormalities will NOT be considered evidence of metastasis
* Patients must have a performance status of 0, 1, or 2; the Lansky performance score should be used for patients < 16 years and the Karnofsky performance score for patients >= 16 years
* Patients who have received prior chemotherapy (excluding steroids) or radiation therapy, except for patients transferring from ARST0331 (low-risk study), are not eligible
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 ml/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * 1 month to < 6 months: 0.4 mg/dL
  * 6 months to < 1 year: 0.5 mg/dL
  * 1 to < 2 years: 0.6 mg/dL
  * 2 to < 6 years: 0.8 mgt/dL
  * 6 to < 10 years: 1 mg/dL
  * 10 to < 13 years: 1.2 mg/dL
  * 13 to < 16 years: 1.5 mg/dL (males) or 1.4 mg/dL (females)
  * >= 16 years: 1.7 mg/dL (males) or 1.4 mg/dL (females)
* Patients with urinary tract obstruction by tumor must meet the renal function criteria AND must have unimpeded urinary flow established via decompression of the obstructed portion of the urinary tract
* Total bilirubin =< 1.5 x upper limit of normal for age
* Peripheral absolute neutrophil count (ANC) >= 750/uL
* Platelet count >= 75,000/uL (transfusion independent)
* No evidence of uncontrolled infection
* Patients must be able to undergo radiation therapy, if necessary, as specified in the protocol
* Female patients of childbearing potential must have a negative pregnancy test
* Female patients who are breast feeding must agree to stop breast feeding
* Sexually active patients of childbearing potential must be willing to use effective contraception during therapy and for at least 1 month after treatment is completed
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Max Age: 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 481 (Actual)
Dates: Start 2006-12-26 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas S Hawkins, Principal Investigator — Children's Oncology Group
Locations (226):
- United States (196):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Harbor-University of California at Los Angeles Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Beaumont Children's Hospital-Royal Oak, Royal Oak, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Winthrop Hospital, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (9):
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Children's Hospital-Brisbane, Herston, Queensland
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (17):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Victoria Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - Centre Hospitalier Universitaire de Quebec, Québec
- Starship Children's Hospital, Grafton, Auckland, New Zealand
- San Jorge Children's Hospital, San Juan, Puerto Rico
- Switzerland (2):
  - Swiss Pediatric Oncology Group - Bern, Bern
  - Swiss Pediatric Oncology Group - Geneva, Geneva

REFERENCES:
- [Derived] Casey DL, Chi YY, Donaldson SS, Hawkins DS, Tian J, Arndt CA, Rodeberg DA, Routh JC, Lautz TB, Gupta AA, Yock TI, Wolden SL. Increased local failure for patients with intermediate-risk rhabdomyosarcoma on ARST0531: A report from the Children's Oncology Group. Cancer. 2019 Sep 15;125(18):3242-3248. doi: 10.1002/cncr.32204. Epub 2019 Jun 7. PMID 31174239
- [Derived] Hawkins DS, Chi YY, Anderson JR, Tian J, Arndt CAS, Bomgaars L, Donaldson SS, Hayes-Jordan A, Mascarenhas L, McCarville MB, McCune JS, McCowage G, Million L, Morris CD, Parham DM, Rodeberg DA, Rudzinski ER, Shnorhavorian M, Spunt SL, Skapek SX, Teot LA, Wolden S, Yock TI, Meyer WH. Addition of Vincristine and Irinotecan to Vincristine, Dactinomycin, and Cyclophosphamide Does Not Improve Outcome for Intermediate-Risk Rhabdomyosarcoma: A Report From the Children's Oncology Group. J Clin Oncol. 2018 Sep 20;36(27):2770-2777. doi: 10.1200/JCO.2018.77.9694. Epub 2018 Aug 9. PMID 30091945
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 481 excludes 33 ineligible cases (declared by the Study Chair) .
Groups:
- Vincristine, Dactinomycin, Cyclophosphamide (VAC): Patients receive VAC chemotherapy comprising vincristine IV over 1 minute on day 1 of weeks 1-13, 16, 19-25, 28, 31-37, and 40; dactinomycin IV over 1-5 minutes on day 1 of weeks 1, 4, 13, 16, 19, 22, 25, 28, 31, 34, 37,and 40; and cyclophosphamide IV over 1 hour on day 1 of weeks 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 31, 34, 37, and 40. Patients may also undergo radiotherapy 5 days a week for 4-6 weeks beginning in week 4.
  Dactinomycin: Given IV Cyclophosphamide: Given IV Vincristine Sulfate: Given IV Radiation Therapy: Undergo radiotherapy Laboratory Biomarker Analysis: Correlative studies Questionnaire Administration: Ancillary studies
- VAC Alternating With Vincristine, Irinotecan (VI): Patients receive VAC chemotherapy alternating with VI chemotherapy comprising vincristine IV over 1 minute on day 1 of weeks 1-13, 16, 17, 19, 20, 22-26, 28, 31-34, 37, 38, and 40; dactinomycin IV over 1-5 minutes on day 1 of weeks 1, 13, 22, 28, 34, and 40; cyclophosphamide IV over 1 hour on day 1 of weeks 1,10, 13, 22, 28, 34, and 40; and irinotecan hydrochloride IV over 1 hour on days 1-5 of weeks 4, 7, 16, 19, 25, 31, and 37. Patients may also undergo radiotherapy 5 days a week for 4-6 weeks beginning in week 4.
Period: Overall Study
Arm/Group | Vincristine, Dactinomycin, Cyclophosphamide (VAC) | VAC Alternating With Vincristine, Irinotecan (VI)
Started | 239 | 242
Completed | 187 | 181
Not Completed | 52 | 61
Not completed — Death | 1 | 1
Not completed — Physician Decision | 8 | 13
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Ineligible | 17 | 16
Not completed — Disease progression or relapse | 15 | 22
Not completed — Adverse Event | 6 | 0
Not completed — Refusal of further therapy | 3 | 8

BASELINE CHARACTERISTICS:
Groups:
- Vincristine, Dactinomycin, Cyclophosphamide (VAC): Patients receive VAC chemotherapy comprising vincristine IV over 1 minute on day 1 of weeks 1-13, 16, 19-25, 28, 31-37, and 40; dactinomycin IV over 1-5 minutes on day 1 of weeks 1, 4, 13, 16, 19, 22, 25, 28, 31, 34, 37,and 40; and cyclophosphamide IV over 1 hour on day 1 of weeks 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 31, 34, 37, and 40. Patients may also undergo radiotherapy 5 days a week for 4-6 weeks beginning in week 4.
- Total: Total of all reporting groups
Arm/Group | Vincristine, Dactinomycin, Cyclophosphamide (VAC) | VAC Alternating With Vincristine, Irinotecan (VI) | Total
Number analyzed (Participants) | 239 | 242 | 481
Age, Continuous [Mean (Standard Deviation); unit: months] | 89.85 (73.39) | 97.86 (82.66) | 93.88 (78.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 113 | 222
  Male | 130 | 129 | 259
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39 | 28 | 67
  Not Hispanic or Latino | 191 | 204 | 395
  Unknown or Not Reported | 9 | 10 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 7 | 7 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 37 | 29 | 66
  White | 165 | 181 | 346
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 28 | 23 | 51

OUTCOME MEASURES:

1. Primary Outcome: Event Free Survival (EFS)
Description: Probability of no relapse, secondary malignancy, or death after 4 year in the study
Time Frame: 4 years
Measure: Number (95% Confidence Interval); unit: Probability
Groups:
- VAC Alternating With Vincristine, Irinotecan (VI): Patients receive VAC chemotherapy alternating with VI chemotherapy comprising vincristine IV over 1 minute on day 1 of weeks 1-13,16, 17, 19, 20, 22-26, 28, 31-34, 37, 38, and 40; dactinomycin IV over 1-5 minutes on day 1 of weeks 1, 13, 22, 28, 34, and 40; cyclophosphamide IV over 1 hour on day 1 of weeks 1,10, 13, 22, 28, 34, and 40; and irinotecan hydrochloride IV over 1 hour on days 1-5 of weeks 4, 7, 16, 19, 25, 31, and 37. Patients may also undergo radiotherapy 5 days a week for 4-6 weeks beginning in week 4.
Arm/Group | Vincristine, Dactinomycin, Cyclophosphamide (VAC) | VAC Alternating With Vincristine, Irinotecan (VI)
Number analyzed (Participants) | 222 | 226
Probability | 0.6255 [0.5575 to 0.6934] | 0.5874 [0.5178 to 0.6569]

2. Primary Outcome: Response Rate (RR)
Description: Proportion of patients with complete or partial response. Complete Response (CR): Complete disappearance of the tumor confirmed at > 4 weeks; Partial Response (PR): At least 64% decrease in volume compared to the baseline; Overall Response (OR) = CR + PR.
Time Frame: Reporting Period 1 (Weeks 1 - 15)
Measure: Number (95% Confidence Interval); unit: Proportion
Groups:
- Vincristine, Dactinomycin, Cyclophosphamide (VAC): Patients receive VAC chemotherapy comprising vincristine IV over 1 minute on day 1 of weeks 1-13, 16, 19-25, 28, 31-37, and 40;dactinomycin IV over 1-5 minutes on day 1 of weeks 1, 4, 13, 16, 19, 22, 25, 28, 31, 34, 37,and 40; and cyclophosphamide IV over 1 hour on day 1 of weeks 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 31, 34, 37, and 40. Patients may also undergo radiotherapy 5 days a week for 4-6 weeks beginning in week 4.
Arm/Group | Vincristine, Dactinomycin, Cyclophosphamide (VAC) | VAC Alternating With Vincristine, Irinotecan (VI)
Number analyzed (Participants) | 222 | 226
Proportion | 0.6667 [0.6047 to 0.7287] | 0.6726 [0.6114 to 0.7337]

3. Primary Outcome: Overall Survival (OS)
Description: Probability of being alive after 4 years in the study.
Time Frame: 4 years
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Vincristine, Dactinomycin, Cyclophosphamide (VAC) | VAC Alternating With Vincristine, Irinotecan (VI)
Number analyzed (Participants) | 222 | 226
Probability | 0.7293 [0.6669 to 0.7917] | 0.7223 [0.6583 to 0.7862]

4. Secondary Outcome: Event Free Survival (EFS) Probability VAC and Early (Week 4) Radiotherapy Compared to Delayed (Week 10) Radiotherapy, Using IRSIV for Historic Comparison
Description: Compare 4-year EFS using eligible participants only to the historical rate of 0.65 with IRSI-V. The 4-year EFS is probability of no relapse, secondary malignancy, or death after 4 years in the study. The Delayed (Week 10) Radiotherapy is from IRSI-V, and the number of participants of IRSI-V is unknown, but we have the rate of 0.65.
Time Frame: 4 years
Population: 17 ineligible participants were excluded.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Vincristine, Dactinomycin, Cyclophosphamide (VAC)
Number analyzed (Participants) | 222
Probability | 0.6255 [0.5575 to 0.6934]

5. Secondary Outcome: Local Failure
Description: Compare 2-year local failure rate to the historical rate of 0.13 with IRSI-V. The Delayed (Week 10) Radiotherapy is from IRSI-V, and the number of participants of IRSI-V is unknown, but we have the rate of 0.13.
Time Frame: 2 years
Population: 17 ineligible participants were excluded.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Vincristine, Dactinomycin, Cyclophosphamide (VAC)
Number analyzed (Participants) | 222
Proportion of participants | 0.1757 [0.1256 to 0.2257]

6. Secondary Outcome: Overall Survival (OS) Probability VAC and Early (Week 4) Radiotherapy Compared to Delayed (Week 10) Radiotherapy, Using IRSIV for Historic Comparison
Description: Compare 4-year OS using eligible participants only to the historical rate of 0.70 with IRSI-V. The 4-year OS is probability of being alive after 4 years in the study. The Delayed (Week 10) Radiotherapy is from IRSI-V, and the number of participants of IRSI-V is unknown, but we have the rate of 0.70.
Time Frame: 4 years
Population: 17 ineligible participants were excluded.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Vincristine, Dactinomycin, Cyclophosphamide (VAC)
Number analyzed (Participants) | 222
Probability | 0.7293 [0.6669 to 0.7917]

7. Secondary Outcome: Incidence of Toxicity
Description: Grade 3 or 4 nausea, diarrhea, dehydration, radiation dermatitis, mucositis due to radiation. Severe and undesirable adverse event is considered as grade 3; Life-threatening or disabling adverse event is grade 4. Grade 4 is worse than grade 3.
Time Frame: Up to 15 weeks
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Vincristine, Dactinomycin, Cyclophosphamide (VAC) | VAC Alternating With Vincristine, Irinotecan (VI)
Number analyzed (Participants) | 222 | 226
Probability | 0.2072 [0.1539 to 0.2605] | 0.3673 [0.3044 to 0.4301]

8. Secondary Outcome: Acute and Late Effects of VAC as Delivered on This Study to D9803 VAC
Description: The toxicity rates will be estimated for each phase and course of treatment, and will be compared to the fixed rates under D9803 using one-sided lower confidence intervals for a single proportion without adjustment for multiple comparisons.
Time Frame: Up to 43 weeks
Population: Number of patients with specific adverse events.
Measure: Number; unit: participants
Groups:
- VAC (Weeks 1-15): Reporting period 1 (acute)
- VAC (Weeks 31 - 43): Reporting period 3 (late)
Arm/Group | VAC (Weeks 1-15) | VAC (Weeks 31 - 43)
Number analyzed (Participants) | 222 | 193
participants
  Anemia | 58 | 54
  Febrile Neutropenia | 30 | 17
  Nausea or Hepatopathy | 6 | 1
  Platelet Count Decreased | 27 | 63
  Vomiting | 9 | 2
Statistical Analysis 1: Comparison: VAC (Weeks 1-15); Compare incidence of Anemia to historical rate of 0.40 from D9803, which is Randomized Study of VCR, Actinomycin-D, and CPM (VAC) vs. VAC alternating with VCR, Topotecan, and CPM (VTC) for Patients with Intermediate Risk RMS. Comparing the incidence of anemia with VAC on ARST0531 to the historical rate of 0.40 with VAC on D9803. The 95% one-sided confidence interval for the incidence of anemia will be calculated and evaluated to see if the interval contains the null rate of 0.40; Test type: Superiority or Other; The incidence of anemia = 0.2613, 95% CI 1-sided [upper limit 0.31]
Statistical Analysis 2: Comparison: VAC (Weeks 1-15); Compare incidence of Nausea or Hepatopathy to historical rate of 0.05 from D9803, which is Randomized Study of VCR, Actinomycin-D, and CPM (VAC) vs. VAC alternating with VCR, Topotecan, and CPM (VTC) for Patients with Intermediate Risk RMS. The 95% one-sided confidence interval for the incidence of nausea or hepatopathy will be calculated and evaluated to see if the interval contains the null rate of 0.05; Test type: Superiority or Other; The incidence of nausea or hepatopathy = 0.0270, 95% CI 1-sided [upper limit 0.0449]
Statistical Analysis 3: Comparison: VAC (Weeks 1-15); Compare incidence of Febrile Neutropenia to historical rate of 0.50 from D9803, which is Randomized Study of VCR, Actinomycin-D, and CPM (VAC) vs. VAC alternating with VCR, Topotecan, and CPM (VTC) for Patients with Intermediate Risk RMS. The 95% one-sided confidence interval for the incidence of febrile neutropenia will be calculated and evaluated to see if the interval contains the null rate of 0.50; Test type: Superiority or Other; The incidence of febrile neutropenia = 0.1351, 95% CI 1-sided [upper limit 0.1729]
Statistical Analysis 4: Comparison: VAC (Weeks 1-15); Compare incidence of Platelet Count Decreased to historical rate of 0.70 from D9803, which is Randomized Study of VCR, Actinomycin-D, and CPM (VAC) vs. VAC alternating with VCR, Topotecan, and CPM (VTC) for Patients with Intermediate Risk RMS. The 95% one-sided confidence interval for the incidence of platelet count decreased will be calculated and evaluated to see if the interval contains the null rate of 0.70; Test type: Superiority or Other; The incidence of platelet count decrease = 0.1216, 95% CI 1-sided [upper limit 0.1577]
Statistical Analysis 5: Comparison: VAC (Weeks 1-15); Compare incidence of Vomiting to historical rate of 0.15 from D9803, which is Randomized Study of VCR, Actinomycin-D, and CPM (VAC) vs. VAC alternating with VCR, Topotecan, and CPM (VTC) for Patients with Intermediate Risk RMS. The 95% one-sided confidence interval for the incidence of vomiting will be calculated and evaluated to see if the interval contains the null rate of 0.15; Test type: Superiority or Other; The incidence of vomiting = 0.0405, 95% CI 1-sided [upper limit 0.0623]
Statistical Analysis 6: Comparison: VAC (Weeks 31 - 43); Compare incidence of Anemia to historical rate of 0.40 from D9803, which is Randomized Study of VCR, Actinomycin-D, and CPM (VAC) vs. VAC alternating with VCR, Topotecan, and CPM (VTC) for Patients with Intermediate Risk RMS. 95% one-sided confidence interval for the incidence of anemia will be calculated and evaluated to see if the interval contains the null rate of 0.40; Test type: Superiority or Other; The incidence of anemia = 0.2798, 95% CI 1-sided [upper limit 0.3329]
Statistical Analysis 7: Comparison: VAC (Weeks 31 - 43); [analysis description as in outcome 8, analysis 2]; Test type: Superiority or Other; The incidence of nausea or hepatopathy = 0.0052, 95% CI 1-sided [upper limit 0.0137]
Statistical Analysis 8: Comparison: VAC (Weeks 31 - 43); [analysis description as in outcome 8, analysis 3]; Test type: Superiority or Other; The incidence of febrile neutropenia = 0.0881, 95% CI 1-sided [upper limit 0.1216]
Statistical Analysis 9: Comparison: VAC (Weeks 31 - 43); [analysis description as in outcome 8, analysis 4]; Test type: Superiority or Other; The incidence of platelet count decrease = 0.3264, 95% CI 1-sided [upper limit 0.3819]
Statistical Analysis 10: Comparison: VAC (Weeks 31 - 43); [analysis description as in outcome 8, analysis 5]; Test type: Superiority or Other; The incidence of vomiting = 0.0104, 95% CI 1-sided [upper limit 0.0224]

9. Secondary Outcome: Compare Event Free Survival (EFS) With Respect to the Level of % Change in FDG PET Maximum Standard Uptake Value (SUVmax) at Week 4
Description: 4-year EFS (probability of no relapse, secondary malignancy, or death after 4 years in the study).
Time Frame: 4 years
Population: 452 participants were excluded due to ineligibility or absence of SUVmax evaluation at baseline and week 4.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | % Change in SUVmax From Baseline to Week 4 < 40% | % Change in SUVmax From Baseline to Week 4 >= 40%
Number analyzed (Participants) | 7 | 22
Probability | 0.2857 [0.0000 to 0.6204] | 0.6364 [0.4354 to 0.8374]

10. Secondary Outcome: Compare Event Free Survival (EFS) With Respect to the Level of % Change in FDG PET Maximum Standard Uptake Value (SUVmax) at Week 15
Description: 4-year EFS (probability of no relapse, secondary malignancy, or death after 4 years in the study)
Time Frame: 4 years
Population: 421 participants were excluded due to ineligibility or absence of SUVmax evaluation at baseline and week 15.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | % Change in SUVmax From Baseline to Week 15 < 40% | % Change in SUVmax From Baseline to Week 15 >= 40%
Number analyzed (Participants) | 9 | 51
Probability | 0.6667 [0.2895 to 1.0000] | 0.5686 [0.4303 to 0.7070]

11. Secondary Outcome: Incidence of Toxicity Related to VI Treatment in Patients With UGT1A1 Genotype
Description: Severe and undesirable adverse event is considered as grade 3; Life-threatening or disabling adverse event is grade 4. Grade 4 is worse than grade 3.
Time Frame: Weeks 4-9 (the first exposure to VI)
Population: Ineligible patients are excluded. Only patients tested for the UGT1A1 genotypes are reported and included in this analysis.
Measure: Number; unit: Counts
Arm/Group | UGT1A1 Genotype 6/6 | UGT1A1 Genotype 6/7 | UGT1A1 Genotype 7/7
Number analyzed (Participants) | 49 | 65 | 12
Counts
  Neutropenia, with or without Fever | 16 | 22 | 4
  Diarrhea | 5 | 14 | 5
Statistical Analysis 1: Comparison: UGT1A1 Genotype 6/6 vs UGT1A1 Genotype 6/7 vs UGT1A1 Genotype 7/7; The incidences of grade 3 or higher neutropenia, with or without fever between UGT1A1 Genotypes (6/6, 6/7, 7/7) were compared by the Fisher's exact test; Test type: Superiority or Other; p = 0.99, Fisher Exact
Statistical Analysis 2: Comparison: UGT1A1 Genotype 6/6 vs UGT1A1 Genotype 6/7 vs UGT1A1 Genotype 7/7; The incidences of grade 3 or higher diarrhea between UGT1A1 Genotypes (6/6, 6/7, 7/7) were compared by Fisher's exact test; Test type: Superiority or Other; p = 0.036, Fisher Exact

12. Secondary Outcome: Toxicity With CYP2B6 Genotypes
Description: Incidence of toxicity related to VAC treatment in patients with CYP2B6 genotypes.
Time Frame: During the study
Population: The analysis was abandoned due to low incidence of toxicity. Data were not collected.
Arm/Group | Vincristine, Dactinomycin, Cyclophosphamide (VAC)
Number analyzed (Participants) | 0

13. Secondary Outcome: Toxicity With GSTA1 and CYP2C9 Genotypes
Description: Incidence of toxicity related to VAC treatment in patients with GSTA1 and CYP2C9 genotypes.
Time Frame: During the study
Population: The analysis was abandoned due to low incidence of toxicity. Data were not collected.
Arm/Group | Vincristine, Dactinomycin, Cyclophosphamide (VAC)
Number analyzed (Participants) | 0

14. Secondary Outcome: Event Free Survival (EFS) by PAX Status
Time Frame: 4 years
Population: Only eligible patients who were tested for their fusion status and PAX partners.
Measure: Number (95% Confidence Interval); unit: Probability
Groups:
- PAX3: Fusion positive with PAX3 partner
- PAX7: Fusion positive with PAX7 partner
Arm/Group | PAX3 | PAX7
Number analyzed (Participants) | 88 | 21
Probability | 0.51 [0.39 to 0.64] | 0.66 [0.37 to 0.94]

15. Secondary Outcome: Incidence of Bladder Dysfunction
Description: Number of patients with a summary score greater than 8.5
Time Frame: 3-6 years after enrollment
Population: 470 participants were excluded due to ineligibility or absence of the dysfunctional voiding and incontinence symptoms questionnaire.
Measure: Number; unit: Participant
Arm/Group | Vincristine, Dactinomycin, Cyclophosphamide (VAC) | VAC Alternating With Vincristine, Irinotecan (VI)
Number analyzed (Participants) | 7 | 4
Participant | 2 | 1

ADVERSE EVENTS:
Description: All eligible patients were considered in the evaluation of adverse events.
Groups:
- VAC Alternating With VI: Patients receive VAC chemotherapy alternating with VI chemotherapy comprising vincristine IV over 1 minute on day 1 of weeks 1-13, 16, 17, 19, 20, 22-26, 28, 31-34, 37, 38, and 40; dactinomycin IV over 1-5 minutes on day 1 of weeks 1, 13, 22, 28, 34, and 40; cyclophosphamide IV over 1 hour on day 1 of weeks 1,10, 13, 22, 28, 34, and 40; and irinotecan hydrochloride IV over 1 hour on days 1-5 of weeks 4, 7, 16, 19, 25, 31, and 37. Patients may also undergo radiotherapy 5 days a week for 4-6 weeks beginning in week 4.
  Irinotecan Hydrochloride: Given IV
  Dactinomycin: Given IV
  Cyclophosphamide: Given IV
  Vincristine Sulfate: Given IV
  Radiation Therapy: Undergo radiotherapy
  Laboratory Biomarker Analysis: Correlative studies
  Questionnaire Administration: Ancillary studies
Arm/Group | Vincristine, Dactinomycin, Cyclophosphamide (VAC) | VAC Alternating With VI
Serious Adverse Events (participants affected / at risk) | 4/222 | 11/226
Other Adverse Events (participants affected / at risk) | 209/222 | 213/226
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vincristine, Dactinomycin, Cyclophosphamide (VAC) (N=222) | VAC Alternating With VI (N=226)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Death NOS (General disorders) | 0 (0) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 3 (3) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vincristine, Dactinomycin, Cyclophosphamide (VAC) (N=222) | VAC Alternating With VI (N=226)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal infection (Infections and infestations) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 9 (11) | 12 (14)
Abducens nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 19 (21) | 16 (22)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Anal mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anaphylaxis (Immune system disorders) | 4 (4) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 102 (183) | 57 (89)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 24 (30) | 35 (42)
Aphonia (Nervous system disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 11 (13) | 7 (8)
Ataxia (Nervous system disorders) | 0 (0) | 3 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Bladder infection (Infections and infestations) | 2 (2) | 3 (3)
Bladder spasm (Renal and urinary disorders) | 1 (1) | 2 (4)
Blood bilirubin increased (Investigations) | 3 (3) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 6 (8) | 13 (15)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 4 (4)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (5) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 10 (10) | 23 (26)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 3 (3)
Dermatitis radiation (Injury, poisoning and procedural complications) | 6 (6) | 2 (2)
Device related infection (Infections and infestations) | 2 (2) | 4 (5)
Diarrhea (Gastrointestinal disorders) | 14 (17) | 51 (63)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (3)
Dysesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Edema trunk (General disorders) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 5 (6) | 10 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Esophageal infection (Infections and infestations) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 3 (4)
External ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Extraocular muscle paresis (Eye disorders) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 3 (3)
Eyelid function disorder (Eye disorders) | 1 (1) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Facial pain (General disorders) | 1 (1) | 3 (3)
Fatigue (General disorders) | 0 (0) | 5 (5)
Febrile neutropenia (Blood and lymphatic system disorders) | 62 (86) | 46 (57)
Fever (General disorders) | 9 (10) | 11 (11)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 2 (2)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0)
GGT increased (Investigations) | 2 (2) | 1 (1)
Gum infection (Infections and infestations) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 4 (6) | 3 (3)
Hearing impaired (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Hematuria (Renal and urinary disorders) | 3 (4) | 1 (1)
Hemoglobin increased (Investigations) | 1 (1) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4) | 11 (14)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 3 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3) | 4 (5)
Hypoglossal nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 24 (25) | 34 (40)
Hyponatremia (Metabolism and nutrition disorders) | 14 (16) | 15 (15)
Hypophosphatemia (Metabolism and nutrition disorders) | 7 (8) | 3 (4)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (7)
Ileus (Gastrointestinal disorders) | 1 (1) | 6 (6)
Infections and infestations - Other, specify (Infections and infestations) | 40 (60) | 37 (56)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (1) | 0 (0)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 2 (2)
Lung infection (Infections and infestations) | 0 (0) | 4 (4)
Lymphocyte count decreased (Investigations) | 48 (144) | 57 (148)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 25 (31) | 46 (48)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (10) | 26 (41)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 2 (2)
Neutrophil count decreased (Investigations) | 179 (484) | 177 (436)
Nystagmus (Nervous system disorders) | 0 (0) | 1 (1)
Oculomotor nerve disorder (Nervous system disorders) | 0 (0) | 2 (4)
Optic nerve disorder (Eye disorders) | 0 (0) | 2 (4)
Oral pain (Gastrointestinal disorders) | 3 (4) | 7 (7)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Pain (General disorders) | 4 (9) | 9 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Penile pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 29 (38) | 26 (44)
Peripheral sensory neuropathy (Nervous system disorders) | 16 (21) | 13 (19)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Platelet count decreased (Investigations) | 94 (164) | 37 (52)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural infection (Infections and infestations) | 1 (1) | 0 (0)
Portal hypertension (Hepatobiliary disorders) | 2 (2) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 1 (1)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Recurrent laryngeal nerve palsy (Nervous system disorders) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Serum amylase increased (Investigations) | 1 (1) | 0 (0)
Sinus pain (Nervous system disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 3 (3) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 5 (5) | 7 (7)
Small intestine infection (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 2 (3)
Thromboembolic event (Vascular disorders) | 1 (1) | 3 (3)
Tracheal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Upper respiratory infection (Infections and infestations) | 3 (4) | 4 (4)
Urethral infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 10 (11) | 8 (13)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Vaginal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vagus nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 16 (17) | 28 (37)
Vulval infection (Infections and infestations) | 1 (1) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 1 (1)
Weight gain (Investigations) | 0 (0) | 2 (3)
Weight loss (Investigations) | 13 (14) | 23 (32)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
White blood cell decreased (Investigations) | 100 (235) | 96 (219)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Wound infection (Infections and infestations) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.